CLINICAL TRIAL: NCT05605626
Title: Operative Vaginal Delivery in Residents and Young Specialists
Brief Title: Learning Skills in Young Specialists and Residents in Operative Vaginal Delivery Using Simulator Models
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Collaborators: Santo Spirito Hospital, Italy (Other)
Responsible Party: Principal Investigator, Claudio Celentano, Clinical Professor, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Other Study IDs: ObGynEASC001
Record Dates: First submitted 2022-03-26; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Birth Disorder; Delivery Complication
Keywords: vaginal birth; vacuum delivery; operative vaginal birth; mannequin training program
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simulator training before: group exposed directly to simulator training without knowing the topic of obstetric emergency
  Interventions: Other: the better retaining of skills
- lesson before simulation training: group undergoing formal lecture before the vacuum delivery simulation on mannequin
  Interventions: Other: the better retaining of skills

INTERVENTIONS:
Other: the better retaining of skills — identify which teaching program has the better retaining of skills

SUMMARY:
Evaluation of different learning programs on persistence of skills in operative vaginal delivery

DETAILED DESCRIPTION:
Investigators enrolled residents and young specialist randomly exposed to simulation of operative vaginal delivery or a lecture before and after experience on simulator program. The two groups were exposed after 8-12 weeks to a second experience of simulator program due to evaluate the improve, deterioration of skills in operative vaginal delivery.

12-months persistence of skills were evaluated

ELIGIBILITY:
Inclusion Criteria: residents or young specialists (less than 5 years after ending of residency) -

Exclusion Criteria: medical students before MD

-

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male/female rate NS in two groups
Study Population: participants were residents in ObGyn or young specialists in ObGyn (less than 5 years)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
improving and retaining skills in two different groups of teaching programs | 12 weeks and 1 year
  evaluate video recorded simulations using items and total value during the operative vaginal delivery on manequin

SECONDARY OUTCOMES:
improve skills in obstetric emergencies considering year of formation and teaching programs | 12 weeks and 1 year
  Comparison of quality scale per items

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chieti, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No
Simulation in EASC

DOCUMENTS (1):
  • Informed Consent Form (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT05605626/ICF_000.pdf